CLINICAL TRIAL: NCT00377299
Title: A Double-blind, Placebo-controlled Pilot Study of Citicoline add-on Therapy in Patients With Bipolar Disorder or Major Depressive Disorder and Amphetamine Abuse or Dependence
Brief Title: A Pilot Study of Citicoline add-on Therapy in Patients With Bipolar Disorder or Major Depressive Disorder and Amphetamine Abuse or Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 052006-27
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-07

CONDITIONS: Amphetamine Abuse; Amphetamine Dependence; Bipolar Disorder; Major Depressive Disorder
Keywords: Amphetamine Abuse; Amphetamine Dependence; Bipolar Disorder; Major Depressive Disorder; Citicoline
MeSH Terms: conditions — Amphetamine-Related Disorders; Bipolar Disorder; Depressive Disorder, Major | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citicoline (Experimental): Citicoline is an over the counter supplement that may have neuroprotective properties and may have antidepressant effects.
  Interventions: Drug: Citicoline
- Placebo (Placebo Comparator): Placebo matching active medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citicoline — Citicoline is an over the counter supplement that may have neuroprotective properties and may have antidepressant effects. Citicoline or placebo (identical in appearance) add-on therapy was given beginning at one tablet (500mg/day) with an increase to two tablets (1000 mg/day) at week 2, three tablets (1500 mg/day) at week 4 and four tablets (2000 mg/day) at week 6. Doses were decreased, if needed, due to side effects.
  Arms: Citicoline
Drug: Placebo — Placebo matching active medication in all other physical aspects
  Arms: Placebo

SUMMARY:
Bipolar disorder (BD) is a common and severe psychiatric illness. Drug and alcohol abuse are very common in people with BD and other mood disorders and are associated with increased rates of hospitalization, violence towards self and others, medication non-adherence and cognitive impairment. However, few studies have investigated the treatment of dual-diagnosis patients as substance use is frequently an exclusion criterion in clinical trials of patients with BD. To address this need, we have developed a research program that explores the pharmacotherapy of people with BD and substance related-disorders. A potentially very interesting treatment for BD is citicoline. Some data suggest that this supplement may stabilize mood, decrease drug use and craving, and improve memory. We found promising results with citicoline in patients with BD and cocaine dependence. In recent years the use of amphetamine and methamphetamine has become an important public health concern. However, virtually no research has been conducted on the treatment of amphetamine abuse. We propose a double-blind placebo controlled prospective trial of citicoline in a group of 60 depressed outpatients with bipolar disorder, depressed phase or major depressive disorder and amphetamine abuse/dependence, to explore the safety and tolerability of citicoline, and its efficacy for mood symptoms, stimulant use and craving and its impact on cognition. Our goal is to determine which symptoms (e.g. mood, cognition, substance use) citicoline appears to be most effective and estimate effect sizes for future work.

DETAILED DESCRIPTION:
Sixty outpatients meeting the inclusion and exclusion criteria will be enrolled after completing an Institutional Review Board (IRB)-approved informed consent process. Baseline evaluation will include a medical and psychiatric history, structured clinical interview for Diagnostic and Statistical Manual (DSM-IV) (SCID), mood assessment with the Inventory of Depressive Symptomatology-Self Report (IDS-C), Young Mania Rating Scale (YMRS), and cognitive assessment with the Hopkins Auditory Verbal Learning Test (HVLT) (similar to the Rey Auditory Verbal Learning Test (RAVLT) but more alternative equivalent versions are available), Stroop and computer assessments including Sternberg Memory Task and the Running Memory Continuous Performance Test. Alternate but equivalent versions of all cognitive tests, except the Stroop, will be used to minimize practice effects with repeated administration. Days and amounts of amphetamine and other substance use will be assessed at each visit with urine drug screens, and through self-report using the timeline follow-back method. Amphetamine, and other drug, craving will be assessed with a visual analogue scales. Citicoline or placebo add-on therapy will be given beginning at one tablet (500mg)/day with an increase to two tablets 1000 mg/day at week 2, three tables 1500 mg/day at week 4 and four tablets 2000 mg/day at week 6.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-70 years
* Meeting criteria for a current major depressive episode (bipolar I,II, not otherwise specified (NOS)

  , depressed phase) or major depressive disorder on the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID) with a duration of at least 4 weeks
* Meeting criteria for amphetamine abuse or dependence with use within 14 days prior to baseline
* No psychotropic medication changes within 14 days prior to study entry

Exclusion Criteria:

* Pregnant or nursing women
* Current citicoline therapy
* Active suicidal or homicidal ideation with plan and intent
* Dementia, mental retardation or other severe cognitive impairment that might interfere with the informed consent process
* Currently incarcerated at a prison or jail
* Severe or life threatening medical condition (e.g. terminal cancer, congestive heart failure)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Psychoneuroendocrine Research Program, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty depressed outpatients with methamphetamine dependence were enrolled and randomized for 12 weeks of acute treatment after completing an IRB-approved written informed consent The study was conducted at the UT Southwestern Medical Center in Dallas. The first participant was enrolled on 10/11/06 and the final assessment was on 4/7/09.
Groups:
- Citicoline: Citicoline add-on therapy was given beginning at one tablet(500mg/day) with an increase to two tablets(1000mg/day) at week 2, three tablets(1500mg/day)at week 4 and four tablets (2000mg/day) at week 6. Patients remained on 2000mg/day throughout the remaining weeks of the study (week 12). Doses were decreased, if needed, due to side effects.
- Placebo: Placebo identical in appearance to the medication was given beginning at one tablet with an increase to two tablets at week 2, three tablets at week 4 and four tablets at week 6. Patients remained on four tables throughout the remaining weeks of the study (week 12). Doses were decreased, if needed, due to side effects.
Period: Overall Study
Arm/Group | Citicoline | Placebo
Started | 32 | 28
Completed | 13 | 4
Not Completed | 19 | 24
Not completed — Lost to Follow-up | 14 | 19
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citicoline | Placebo | Total
Number analyzed (Participants) | 32 | 28 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 41.0 (9.6) | 34.0 (7.4) | 37.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 20 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Depression Symptoms
Description: Inventory of Depressive Symptomatology-Clinician Rated (IDS-C), (a clinician-administered depression scale) is used to assess the severity of depressive symptoms.Scores can range from 0 to 84. The higher the score, the worse the depressive symptoms(worse outcome).
Time Frame: 12 weeks
Population: The intent to treat (ITT) group includes all who returned for at least one post baseline visit. Analysis uses Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Placebo: Placebo.
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 28 | 20
scores on a scale | 26.2 (2.5) | 33.1 (3.0)
Statistical Analysis 1: Comparison: Citicoline vs Placebo; Test type: Superiority or Other; p = 0.05, ANCOVA — Significance was set at a p value of ≤ 0.05

2. Secondary Outcome: Amphetamine Craving
Description: Visual Analog Scale (VAS) assessing Methamphetamine craving with a 1-100 scale.Higher values on the VAS scale indicate a higher Methamphetamine craving(worse outcome).
Time Frame: 12 Weeks
Population: ITT includes those returning for at least one post baseline visit. LOCF used for end point data.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 19 | 27
scores on a scale | 31.9 (8.0) | 44.1 (9.7)
Statistical Analysis 1: Comparison: Citicoline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA — Significance was set at a p value of ≤ 0.05

3. Secondary Outcome: Amphetamine Use
Description: Participant reported days per 7-day week of methamphetamine use.
Time Frame: 12 weeks
Population: ITT includes those returning for at least one post baseline visit. LOCF used for end point data.
Measure: Mean (Standard Error); unit: days per week
Groups:
- Placebo: Placebo matching Citicoline.
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 28 | 20
days per week | 2.9 (0.6) | 2.3 (0.5)
Statistical Analysis 1: Comparison: Citicoline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA — Significance was set at a p value of ≤ 0.05

4. Secondary Outcome: Hopkins Auditory Verbal Learning Test (HVLT)
Description: The Hopkins Auditory Verbal Learning Test (HVLT) is a measure of cognition (memory/recall). Raw scores are derived for Total Recall, Delayed Recall, Retention (% retained), and a Recognition Discrimination Index. Raw scores are calculated into T-scores. T-scores are standardized scores on each dimension for each type. A score of 50 represents the mean. A difference of 10 from the mean indicates a difference of one standard deviation. Thus, a score of 60 is one standard deviation above the mean, while a score of 30 is two standard deviations below the mean.
Time Frame: 12 weeks
Population: ITT includes those returning for at least one post baseline visit. LOCF used for end point data.
Measure: Mean (Standard Error); unit: T score
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 17 | 9
T score | 38.5 (3.8) | 47.5 (4.7)
Statistical Analysis 1: Comparison: Citicoline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA — Significance was set at a p value of ≤ 0.05

5. Secondary Outcome: Stroop Color Word Test
Description: The Stroop Color Word Test measures the individual's ability to separate the word and color naming stimuli thus the ability to sort information from the environment and selectively react to this information. The scoring is a measure of time to complete 100 items and the numbers of items that can be completed. THe scores are converted into T-scores which have a mean of 50 and a standard deviation of 10.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: T score
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 28 | 20
T score | 56.2 (2.6) | 54.3 (3.1)
Statistical Analysis 1: Comparison: Citicoline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA — Significance was set at a p value of ≤ 0.05

ADVERSE EVENTS:
Arm/Group | Citicoline | Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 4/28
Other Adverse Events (participants affected / at risk) | 2/32 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citicoline (N=32) | Placebo (N=28)
Injuries Due to Car Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant was in a motor vehicle accident.
Drug Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Overdose.
Drug Overdose / Suicidal Gesture (Psychiatric disorders) | 0 (0) | 1 (1) — Overdose.
Car Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant was in a motor vehicle accident.
Psychiatric Hospitalization Involuntary (Psychiatric disorders) | 0 (0) | 1 (1) — Psychiatric hospitalization.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citicoline (N=32) | Placebo (N=28)
Severe Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) — Participant with a history of panic attacks experienced a severe panic attack. Attack resolved without need for medical intervention.
Tooth Abscess and Infection (Infections and infestations) | 1 (1) | 0 (0) — Participant reported an abscessed/infected tooth and received amoxycillin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes